CLINICAL TRIAL: NCT00415779
Title: Phase I Study of the Combination of Zoledronic Acid and Docetaxel in Patients With Hormone Refractory Metastatic Prostate Cancer
Brief Title: ZANTE: Zometa and Taxotere in Hormone Refractory Prostate Cancer
Acronym: ZANTE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Francesco Perrone, Director Clinical Trials Unit, National Cancer Institute Naples, Italy
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZANTE; EUDRACT 2006-000426-31
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Metastatic Prostate Cancer
Keywords: hormone refractory; bone metastasis; chemotherapy; biphosphonates
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: docetaxel — given IV in subsequent cohorts of patients at 30, 40, or 50mg/m2
Drug: zoledronic acid — 2 mg IV every 2 weeks

SUMMARY:
This phase I trial is studying the side effects and best dose of docetaxel when given with zoledronic acid in patients with bone metastasis from prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
Docetaxel has been used alone and in combination with other anti-cancer therapies in the treatment of hormone refractory metastatic prostate cancer. Zoledronic acid has been used in the treatment of bone metastasis from prostate cancer. This is a study of the combination of these two agents. The Zante study will test a dose escalation of docetaxel in association with a predetermined dose of zoledronic acid (2 mg), given every 14 days for a minimum of 6 and maximum of 12 cycles.

Sequence A: Docetaxel on day 1 and zoledronic acid on day 2

Sequence B: Zoledronic acid on day 1 and docetaxel on day 2

Patients are enrolled sequentially in cohorts of 3 for each dose level, and a maximum of 36 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Hormone refractory prostate cancer
* Stage IV disease with bone metastasis
* No immunotherapy, hormonal therapy or radiotherapy within the previous month
* Performance status < or = 2 (ECOG)
* Serum creatinine < 1.5 mg/100ml
* Serum bilirubin < or = 1.25 x UNL (upper normal limit) (or < or = 1.5 x UNL in the presence of hepatic metastases); SGOT e SGPT < or = 1.5 x UNL (or < or = 2.5 x UNL in presence of hepatic metastases)
* Left ventricular ejection fraction > or = 50% (measured by cardiac ultrasound or MUGA scan)
* Neutrophils > 1500/mm3; platelets >100000/mm3; hemoglobin >10 g/100 ml· Life expectancy of at least 3 months

Exclusion Criteria:

* Previous malignancies with the exception of radically treated epithelioma
* Previous chemotherapy
* Comorbidities that would, in the Investigator's opinion, contraindicate the use of the drugs in the study
* Uncontrolled Diabetes
* Severe cardiac arrhythmias, severe uncontrolled congestive heart failure, severe ischemic cardiac disease or myocardial infarction within the previous 6 months
* severe infection
* cerebral metastasis
* Pre-existing motor or sensory neurotoxicity > or = grade 2 according to CTC (Common Toxicity Criteria).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-12 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
to determine the maximum tolerated dose and dose limiting toxicity of docetaxel in the two treatment schedules | every 2 weeks for up to 3 cycles

SECONDARY OUTCOMES:
to determine the recommended docetaxel dose when combined with zoledronic acid for phase II studies | every 2 weeks for 6 cycles
to determine which administration sequence of the combination permits a higher dosage of docetaxel | every 2 weeks for 6 weeks
to describe the toxicity of the combination of the two drugs | every 2 weeks
to describe the effects of the combination of the two drugs on biologic parameters: angiogenetic factors, cytokines, differential neuroendocrine markers, serum markers of osteolysis | every 12 weeks
to describe the antitumor activity of the two drug association | every 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michele Caraglia, M.D., Principal Investigator — Experimental Pharmacology, National Cancer Institute Naples; Alfredo Budillon, M.D., Principal Investigator — Experimental Pharmacology, National Cancer Institute Naples; Francesco Perrone, M.D., Ph.D, Principal Investigator — National Cancer Institute Naples, Italy; Director Clinical Trials Unit; R. Vincenzo Iaffaioli, M.D, Principal Investigator — Medical Oncology B, National Cancer Institute Naples; Gaetano Facchini, M.D., Principal Investigator — Medical Oncology B, National Cancer Institute Naples; Alessandro Morabito, M.D., Principal Investigator — Clinical Trials Unit, National Cancer Institute Naples
Locations (2):
- Italy (2):
  - Istituto Nazionale dei Tumori, Napoli
  - Ospedale Oncologico Regionale C.R.O.B. - Basilicata, Rionero in Vulture